CLINICAL TRIAL: NCT00124371
Title: Fit For Surgery Study: A Randomised Controlled Trial of a Nurse-Led Programme to Optimise Mental and Physical Fitness for Surgery and Coronary Risk Factor Control in Patients Waiting for Coronary Artery Bypass Surgery
Brief Title: Programme to Optimise Risk Factors in Patients Waiting for Coronary Artery Bypass Surgery
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Royal Brompton & Harefield NHS Foundation Trust (Other)
Collaborators: British Heart Foundation (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2001HS030B; DHSAEPC2675; 01-180; PG02/116/14483
Record Dates: First submitted 2005-07-25; First posted 2005-07-27 (Estimated); Last update posted 2005-08-05 (Estimated); Status verified 2005-07

CONDITIONS: Coronary Artery Disease
Keywords: coronary artery bypass surgery; risk factors; nurse-led secondary prevention; prehabilitation; waiting period
MeSH Terms: conditions — Coronary Artery Disease

INTERVENTIONS:
Behavioral: a nurse led home-based education and support programme

SUMMARY:
The time spent waiting for heart surgery can be extremely stressful. This programme aims to address this by providing a home-based, nurse-led support and education programme. Patients will be followed up in their own homes monthly by a cardiac nurse and given lifestyle advice and information to prepare them for surgery. This will be evaluated to test whether providing this support improves patients' anxiety and quality of life while they wait and also whether their blood pressure, weight and cholesterol are reduced and they have a smoother recovery as a consequence.

DETAILED DESCRIPTION:
While waiting for coronary artery bypass graft (CABG) surgery many patients receive little if any medical and nursing input, at a time which is very stressful for them and their families. This randomised controlled trial will test whether a home-based, nurse-led support and education programme for patients waiting for such surgery can optimise mental and physical fitness and improve coronary heart disease risk factors by addressing anxiety, hypertension, obesity, diabetes and serum cholesterol in the waiting period. Patients will be followed up in their own homes monthly by a cardiac nurse and given lifestyle advice and information to prepare them for surgery. Primary outcome measurements will be anxiety, length of stay, blood pressure, cholesterol, blood glucose, smoking and body mass index. Secondary outcomes will be quality of life, and post-operative complications. Economic analysis and qualitative assessment of patients' opinion of the programme will also be performed.

ELIGIBILITY:
Inclusion Criteria:

* Patients waiting for first time cardiac bypass surgery
* Able to read and understand English

Exclusion Criteria:

* Patients living outside designated geographical area (>1.5 hours drive from hospitals)
* Patients having surgery other than first time coronary artery bypass grafts
* Patients unable to read and understand English
* Patients with life-threatening significant non-cardiovascular disease e.g. cancer
* All risk factors under control (blood pressure <140 systolic and/or < 90 diastolic and/or serum cholesterol <5 mmol/L and/or blood glucose < 7mmol/L and anxiety score < 8 on the Hospital Anxiety and Depression Scale).

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200
Dates: Start 2003-01; Study Completion 2005-10

PRIMARY OUTCOMES:
Anxiety
Length of hospital stay
Changes to blood pressure, smoking rate, serum cholesterol, body mass index and blood glucose from baseline

SECONDARY OUTCOMES:
Quality of life
Post-operative complications (cerebrovascular accident [CVA], myocardial infarction [MI], infection (wound & chest), arrhythmia requiring either formal resuscitation, pharmacological intervention or pacing)
Patients' perspective of the impact of the programme on their support and information needs (qualitative interview)

CONTACTS AND LOCATIONS:
Overall Officials: John Pepper, FRCS MChir, Principal Investigator — Royal Brompton and Harefield Hospitals
Locations (1):
- Royal Brompton and Harefield NHS Trust, London, London, United Kingdom

REFERENCES:
- [Background] Goodman H, Peters E, Matthews R, Geraghty A, Godden J, Shuldham C. A pilot study using a newly devised manual in a programme of education and support for patients waiting for coronary artery bypass surgery. Eur J Cardiovasc Nurs. 2003 Apr;2(1):27-37. doi: 10.1016/S1474-5151(02)00044-0. PMID 14622646